CLINICAL TRIAL: NCT04733365
Title: Nursing Rehabilitation on Patients Admitted by Recently Decompensated Heart Failure (ERIC Program) - Impact of Exercise
Brief Title: Exercise in Patients Admitted With Recently Decompensated Heart Failure
Acronym: ERIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Bruno Miguel Delgado, Nurse, Centro Hospitalar do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016.172
Record Dates: First submitted 2017-11-13; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Decompensated Heart Failure; Functional Cardiac Disorder
Keywords: Exercise; Nursing rehabilitation; Functional capacity; Heart failure
MeSH Terms: conditions — Motor Activity; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Patients admitted due to decompensated heart failure who will perform the training protocol - ERIC protocol
  Interventions: Other: ERIC protocol
- Control group (No Intervention): Patients admitted due to decompensated heart failure who will perform the standard rehabilitation nursing care for this type of patients

INTERVENTIONS:
Other: ERIC protocol — ERIC protocol is an aerobic exercise protocol with 5 levels of intensity
  Arms: Training group

SUMMARY:
An aerobic physical exercise protocol will be applied to patients admitted in ward due to decompensated heart failure, in order to validate the efficacy and safety of physical exercise in this phase of clinical stabilization, through the said training protocol - ERIC program.

DETAILED DESCRIPTION:
With the objective of validating the efficacy and safety of physical exercise as a therapeutic resource in patients admitted for decompensated heart failure; will be applied, by rehabilitation nurses, a protocol of physical exercise, with increasing levels of intensity. Patients who meet the inclusion criteria will be randomized through an online program (randomizer.org) and the ERIC protocol will be applied to the test group. The control group will be implemented the usual care of rehabilitation nursing. The ERIC protocol comprises 5 levels of intensity, as following shown:

Stage 1 - respiratory and calisthenic exercises (5-10 minutes) Stage 2 - pedaler for 5-10 minutes Stage 3 - aerobic training: walking on the corridor for 5-10 minutes Stage 4 - aerobic training: walking on the corridor for 10-15 minutes Stage 5 - aerobic training: walking on the corridor for 15 minutes + climbing stairs for 5 minutes

All patients will be monitored and followed up by a rehabilitation nurse while they are doing the exercise. The investigator decides, depending on the patient's performance and clinical conditions, the form of progression in the program, but it is mandatory to follow the previously defined levels of intensity. Patients in the test group may start the program only on stage I or II according to clinical criteria.

At admission of the patients (test group and control group) clinical and sociodemographic parameters are evaluated, as well as data related to Barthel's indices and London Chest of activities of daily living (LCADL). At the discharge date, the Barthel index and the LCADL scale will also be evaluated, as well as the 6-minute walking test.

ELIGIBILITY:
Inclusion Criteria:

* Admission diagnosis of Decompensated heart failure
* More than 18 years old
* Capacity to provide informed consent

Exclusion Criteria:

* Osteoarticular pathology that impedes the performance of the exercise;
* Existence of inotropic infusions;
* Dysrhythmia or precordial pain in the last 24 hours,
* Acute pulmonary edema in the last 12 hours,
* SBP greater than 180mmHg or less than 80 mmHg (except in cases where this is the baseline value for the patient),
* Need for oxygen at a rate greater than 3 l / min,
* Glycemic decompensation in the last 12 hours,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
6 minute walking test | Through study completion, an average of 1 year
  Number of meters walked in the 6 minute walking test

SECONDARY OUTCOMES:
Barthel Index score | Through study completion, an average of 1 yeare
  Barthel evaluates dependence on self-care, it ranges from 0 to 100. The higher score inidcates more independence on the performance of self-care activities
London Chest Activity of Daily Living scale score | Through study completion, an average of 1 year
  LCADL acesses how dyspnea affects self-care. It ranges from 9 to 45, the lower scores represents less dyspnea during the activities, representing a better status.
Cardiac adverse events | Through study completion, an average of 1 year
  Number of adverse events occured during in the training group

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Delgado, MsC, Principal Investigator — Centro Hospitalar do Porto
Locations (3):
- Portugal (3):
  - Hospital Infante D Pedro, Aveiro
  - Hospital Pulido Valente, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia